CLINICAL TRIAL: NCT06155045
Title: A Comparative Study Between Conventional & Modified Carbo-dissection Techniques for LIMA Harvesting in CABG Patients
Brief Title: Comparing a New Technique of Combining Carbon-dioxide With Electrocautery With Usual Technique of Stand-alone Electrocautery for Taking Down Left Internal Mammary Artery for Coronary Artery Bypass(CABG)
Acronym: CABG
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Government Medical College Kottayam (Other)
Responsible Party: Principal Investigator, Dinesh Kumar Sathanantham, Resident in Dept. of Cardiovascular and Thoracic Surgery, Government Medical College Kottayam
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 95/2020
Record Dates: First submitted 2023-11-24; First posted 2023-12-04 (Actual); Last update posted 2023-12-15 (Actual); Status verified 2023-12

CONDITIONS: Coronary Artery Disease; Coronary Artery Disease With Myocardial Infarction
Keywords: CABG, LIMA harvesting, CAD
MeSH Terms: conditions — Coronary Artery Disease; Coronary Artery Disease, Autosomal Dominant, 1

STUDY DESIGN:
Intervention Model Description: The interventional group was compared with the conventional group in terms of two parameters : 1) operative time 2) blood flow/min
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Modified Carbo-dissection technique (Experimental): The carbo-dissection technique is performed using an improvised instrument that combines an electrocautery pencil (ValleylabTM Force FX electrocautery Pencil, Covidien, USA) with a CO2 mister blower (PerfX® Heart Lung pack Blower/Mister Kit, B L Lifesciences, Noida, India) and the instruments are fixed together using silk ties.The electrocautery is used in the coagulation mode at a setting of 10 to 15. The C02 flow is set at 2 to 3 litres/minute. Saline flow is adjusted to a level that does not hinder the effective coagulation but still prevents drying and desiccation of the tissues. Following the dissection of LIMA by the techniques mentioned above, blood flow from the harvested LIMA for one whole minute was noted(1 min post division of LIMA). The operative time required for LIMA dissection was also noted and entered. Patient's s demographic data were also collected and entered.
  Interventions: Procedure: Modified Carbo-dissection Technique
- Conventional Arm (Active Comparator): The conventional technique is performed using an electrocautery pencil (ValleylabTM Force FX electrocautery Pencil, Covidien, USA). The electrocautery is used in the coagulation mode at a setting of 10 to 15. Following the dissection of LIMA, blood flow from the harvested LIMA for one whole minute was noted(1 min post division of LIMA). The operative time required for LIMA dissection was also noted and entered. Patient's s demographic data were also collected and entered.
  Interventions: Procedure: Conventional Arm

INTERVENTIONS:
Procedure: Modified Carbo-dissection Technique — This technique comes the C02 blower with electrocautery. Thereby, producing vasodilatation due to the gas and dissection aided by the electrocautery.
  Arms: Modified Carbo-dissection technique
Procedure: Conventional Arm — This technique uses only the electrocautery as conventional model
  Arms: Conventional Arm

SUMMARY:
The goal of this study is to compare the efficacy of a new harvesting technique for an arterial conduit(LIMA - Left Internal Mammary artery) in patients undergoing Coronary artery bypass grafting. The researcher will compare the

1. Time taken to harvest the artery
2. Flow of blood between the two techniques

DETAILED DESCRIPTION:
Following consultation to our department, after a detailed history and clinical examination,patients with CAD, being planned for CABG, will be subjected to a detailed pre-op Echocardiogram and coronary angiogram. After necessary pre-op assessment, patient will be taken up for the surgery. Invasive monitoring will be done.

Following dissection of LIMA by the above mentioned technique, flow of blood from the harvested LIMA, for one whole minute is noted. The operative time required for the dissection of LIMA will be noted and entered.

The data between the two techniques will be compared statistically.

ELIGIBILITY:
Inclusion Criteria:

1. Elective CABG
2. Hemodynamically stable CAD patients

Exclusion Criteria:

1. Re-operation, previous sternotomy (where LIMA is already dissected)
2. concomitant valve operation, ventricular aneurysm resection
3. other additional major cardiac procedures
4. Patients with chronic obstructive pulmonary disease

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 46 (Actual)
Dates: Start 2021-01-01 (Actual); Primary Completion 2021-12-31 (Actual); Study Completion 2021-12-31 (Actual)

PRIMARY OUTCOMES:
Operative time | 10-20 min
  Time taken to perform the harvesting of the LIMA
Blood flow/min | 1 min
  Post dividing of the LIMA: blood from the LIMA is measured for 1 min

CONTACTS AND LOCATIONS:
Overall Officials: Dinesh Kumar Sathanantham, MBBS MS MCh, Principal Investigator — Government Medical College Kottayam
Locations (1):
- Government Medical College Kottayam, Kottayam, Kerala, India

IPD SHARING:
Plan to Share IPD: No
The two parameters: Operative time and Blood flow/min between two techniques will be shared.
  Co-morbidities data will also be shared

REFERENCES:
- [Background] Gilbert S, Singh D, Sivakumar MK. Modified carbodissection: A new technique for harvesting the internal mammary artery. Multimed Man Cardiothorac Surg. 2017 Oct 29;2017. doi: 10.1510/mmcts.2017.018. PMID 29300076
- [Background] Ozkan M, Koramaz I, Ulus AT, Tavil Y, Filizlioglu H, Baykan EC, Eryilmaz S, Inan B, Katircioglu SF, Ozyurda U. Effect of carbon dioxide insufflation on free internal thoracic artery flows: is it a vasodilator? J Thorac Cardiovasc Surg. 2004 Sep;128(3):354-6. doi: 10.1016/j.jtcvs.2003.11.006. PMID 15354091
- [Result] Lee ME. Carbodissection of the internal thoracic artery pedicle. Ann Thorac Surg. 1988 Oct;46(4):470-1. doi: 10.1016/s0003-4975(10)64671-1. PMID 3140750
- [Derived] Nair JTK, Sathanantham DK, Thomas JK. Comparison of conventional and modified carbo-dissection techniques for LIMA harvesting in CABG. Indian J Thorac Cardiovasc Surg. 2025 Feb;41(2):162-166. doi: 10.1007/s12055-024-01780-z. Epub 2024 Jul 15. PMID 39822879

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-11-11): https://cdn.clinicaltrials.gov/large-docs/45/NCT06155045/Prot_SAP_000.pdf